CLINICAL TRIAL: NCT05585242
Title: Randomized Control Trial of Acceptance and Commitment Therapy Adapted for Women With Infertility-related Distress
Brief Title: Acceptance and Commitment Therapy (ACT) Adapted for Women With Infertility-related Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Principal Investigator, Jennifer Gordon, Principal Investigator, University of Regina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB 2022-026
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2023-04

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized either to the ACT conditions or to the waitlist control condition. Randomization will occur using a 1:1 allocation ratio and random block sizes to ensure comparable condition sizes while minimizing the ability to predict condition assignment.
Masking Description: Blinding will not be implemented as condition assignment through randomization will be obvious to both the participants and the primary investigator. Participants will be provided with an introduction and rationale for the respective condition they are assigned to. Participants in the waitlist control condition will be given the opportunity to enroll in the intervention after completing the follow-up measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The program consists of brief weekly videos, each addressing a particular Acceptance and Commitment Therapy technique to be implemented that week. Participants receive the videos by email from the researcher and watch them on their own. Each video also assigns a "homework" exercise for the participant to complete that week and includes a summary of the module.
  Interventions: Behavioral: Infertility ACTion Program
- Waistlist (No Intervention): Participants in the waitlist control condition will complete the same measures as the intervention group. After they have completed their one-month follow-up measures they will be given the opportunity to receive the intervention.

INTERVENTIONS:
Behavioral: Infertility ACTion Program — Seven 15-minutes videos of Acceptance and commitment therapy adapted for women with infertility with assigned homework and summaries of the videos.
  Arms: Intervention

SUMMARY:
This RCT will test the effect of a 7-week self-help ACT-based program in improving fertility-related quality of life and psychological flexibility, in women with infertility.

DETAILED DESCRIPTION:
Ninety women with infertility living in Canada and the United States will be recruited. They will be emailed seven weekly 15-minute videos, each providing instructions on a new Acceptance and Commitment Therapy-based technique that addresses the impact of infertility on psychological inflexibility and distress. Fertility-related quality of life and psychological flexibility will be measured before and after the program. Outcomes will also be measured at one-month follow-up. Feedback about how to improve the program will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Has been trying to get pregnant for 12+ months and has failed OR is currently undergoing fertility treatments
* Lives in Canada or the United States
* Reports a high level of distress related to infertility, as indicated by a FertiQoL score below 71

Exclusion Criteria:

* Is currently experiencing active suicidal ideation, as indicated by a score of 7 or above on the Suicide Behaviours Questionnaire - Revised (SBQ-R)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Fertility Quality of Life tool (Fertiqol) | Pre-to-post intervention change and in the month following the intervention (post measures assessed 4 weeks after receipt of last module)
  Pre-to-post change in quality of life related to a diagnosis of infertility. Scores range from 0-100, with higher scores indicating better quality of life.
Psychological flexibility (MPFI) | Pre-to-post intervention change and in the month following the intervention (post measures assessed 4 weeks after receipt of last module)
  Pre-to-post change in psychological flexibility. Higher scores on the flexibility sub scale indicating better psychological flexibility.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Pre-to-post intervention change and in the month following the intervention (post measures assessed 4 weeks after receipt of last module)
  Pre-to-post change in anxious symptoms; Scores range from 0-21, with higher scoresindicating more severe anxiety
Patient Health Questionnaire-9 (PHQ-9) | Pre-to-post intervention change and in the month following the intervention (post measures assessed 4 weeks after receipt of last module)
  Pre-to-post change in depressive symptoms; Scores range from 0-27, with higherscores indicating more severe depressive symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No